CLINICAL TRIAL: NCT05665660
Title: Developing and Evaluating Scalable and Culturally Relevant Interventions to Improve Breast Cancer Screening Among White Mountain Apache Women
Brief Title: Developing and Evaluating Culturally Relevant Interventions to Improve Breast Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Native American Research Center for Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: IRB00022667
Record Dates: First submitted 2022-12-19; First posted 2022-12-27 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: mammography; cancer screening
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Women randomized to receive CARE who have not received a mammography at 3 months will be offered CARE+COACH to facilitate completion of their screening and contacted at 4 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARE - Intervention arm for mammography education (Experimental): CARE is a culturally tailored mammography education module.
  Interventions: Behavioral: CARE
- CARE + COACH - Intervention arm for mammography education + a patient navigator (Experimental): CARE + COACH is the CARE education module in addition to a COACH, which is access to an Apache paraprofessional women's health coach. The Coach functions like a patient navigator.
  Interventions: Behavioral: CARE + COACH

INTERVENTIONS:
Behavioral: CARE — CARE is a culturally tailored mammography education module.
  Arms: CARE - Intervention arm for mammography education
Behavioral: CARE + COACH — CARE + COACH is a culturally tailored mammography education module + access to an Apache paraprofessional women's health coach who functions as a patient navigator
  Arms: CARE + COACH - Intervention arm for mammography education + a patient navigator

SUMMARY:
The goal of this study is to evaluate the relative benefits of an intervention to promote breast cancer screening among women in the White Mountain Apache (WMA) community. Women will be randomized to receive CARE, a culturally tailored mammography education module, or CARE+COACH, which is the CARE education module plus access to an Apache paraprofessional women's health coach (i.e., patient navigator). The CARE intervention was developed through a community-based participatory research process. The primary outcome is mammography uptake within 2 months of a referral.

ELIGIBILITY:
Inclusion Criteria:

* Referral for screening mammography from a Whiteriver Indian Health Service provider
* Self-identify as American Indian or Alaska Native (AIAN)
* Female
* Live on within 60 miles of the Fort Apache Indian Reservation

Exclusion Criteria:

* Women who have received a mammogram within the prior 12 months
* Women with a personal history of breast cancer
* Unable to participate in full intervention or evaluation due to an anticipated event (e.g., planned move)
* Unwilling to be randomized

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 323 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Mammography uptake | 2 months
  Mammography uptake within 2 months of referral

CONTACTS AND LOCATIONS:
Overall Officials: Allison Barlow, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Indigenous Health, Whiteriver, Arizona, United States